CLINICAL TRIAL: NCT02277314
Title: Manual Small Incision Cataract Surgery Outcomes in an Educational Setting
Acronym: MSICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Joseph Miller, Joseph Miller, MD, MPH, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1404277367
Record Dates: First submitted 2014-10-24; First posted 2014-10-29 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low Cost Treatment for Cataracts (Other): Low cost, manual small incision cataract surgery performed in an educational environment. All costs covered by subjects.
  Interventions: Procedure: Manual Small Incision Cataract Surgery

INTERVENTIONS:
Procedure: Manual Small Incision Cataract Surgery — This cost-effective solution for removing cataracts, also known as Manual Small Incision Cataract Surgery (MSICS), is a positive alternative when Phaco is not an option due to costs. The procedure takes approximately 30 minutes and involves a mid-size incision and an intraocular lens (IOL), or artificial lens, replacing the natural lens. Following the procedure, patients may need glasses, and most will need bifocals, but overall vision will be significantly improved.
  Other Names: MSICS

SUMMARY:
The overall objective is to determine the visual outcomes and cost to perform Manual Small Incision Cataract Surgery (MSICS) in a small cohort at an academic medical center in the United States. The primary outcome measure will be the percentage of the study group achieving a post operative visual acuity 20/40 Snellen. This percentage will be compared to historical cohorts reported for phacoemulsification cataract surgery (PCS), when performed in academic centers. A secondary outcome will be to determine the actual institutional cost of providing MSICS in the setting of an academic medical center. The hypothesis is that MSICS is appropriate for a teaching environment (as evidenced by a comparable rate of 20/40 acuity or better at 90 days post op, as compared to PCS), and can be provided at a cost that makes visual rehabilitation affordable to the uninsured and underinsured.

DETAILED DESCRIPTION:
The investigator will perform a study of a pilot implementation of portions of the Aravind method of promoting access to care and provision of surgical services in the setting of an academic medical center teaching program. Target enrollment is 100 subjects having cataracts. Potential subjects will be identified through vision screening programs and if cataracts are found they will be offered MSICS at a price deemed to be affordable by individuals without insurance.

A survey of Pima County providers found that $3500 was the lowest price offered to a self-pay patient for one-stage cataract extraction (CPT 66984) for PCS facility fee, surgeon fee, and anesthesia fee. The expectation is that MSICS can be delivered in a teaching environment at a cost of $500. The investigator wishes to determine if this price point is sustainable and if a continuing model of cataract visual rehabilitation service delivery can be safely, affordably, and ethically delivered to those who cannot afford to pay, while integrating resident education and autonomy into the delivery model.

The proposed outcome measure is the proportion of eyes that see 20/40 or better while wearing glasses for those participants that do not have comorbid conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years or older (adults).
2. Medically Stable, able to safely undergo surgery.
3. Nuclear sclerotic cataract
4. Preoperative best corrected visual acuity (BCVA) 20/80 or worse
5. Expected post-operative potential acuity of 20/40 or better
6. Able to pay the $500 cost of surgery at the time of surgery

Exclusion Criteria:

Potential subjects not satisfying any of the above

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Manual Small Incision Cataract Surgery with outcomes of 20/40 or better at the end of a year and with spectacle correction | 2 years
  Post-cataract surgery the subject must have a visual acuity of 20/40 or better with spectacle correction

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Miller, MD, PhD, Principal Investigator — University of Arizona Department of Ophthalmology
Locations (1):
- University of Arizona Medical Center Alvernon Physician Offices, Tucson, Arizona, United States